CLINICAL TRIAL: NCT01126814
Title: A Phase I-II Study Evaluating the Safety and Efficacy of Imatinib Mesylate (Gleevec) Combined With Reinduction Chemotherapy Using Mitoxantrone, Etoposide and Cytarabine in Patients With Relapsed/Refractory C-kit Positive Acute Myeloid Leukemia
Brief Title: A Study of Imatinib With Reinduction Chemotherapy Using Mitoxantrone, Etoposide and Cytarabine in Patients With Relapsed/Refractory C-kit Positive (AML) Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-0147-C
Record Dates: First submitted 2010-05-03; First posted 2010-05-20 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Leukemia
Keywords: Gleevec; c-kit; aml
MeSH Terms: conditions — Leukemia; Piebaldism; Leukemia, Myeloid, Acute | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one (Experimental)
  Interventions: Drug: Imatinib (Gleevec)

INTERVENTIONS:
Drug: Imatinib (Gleevec)

SUMMARY:
This is a Phase I-II study evaluating the toxicity and efficacy of imatinib combined with mitoxantrone, etoposide and high-dose cytarabine reinduction therapy in relapsed and refractory AML. Patients will be treated initially at a 200 mg dose of imatinib; if tolerated, the imatinib dose will be escalated in subsequent cohorts to 300 mg and 400 mg. Once the recommended dose is determined, the remaining patients will be treated at that dose, to evaluate the antileukemic activity of the regimen. Patients achieving complete remission will receive consolidation therapy with imatinib combined with high-dose cytarabine and mitoxantrone, followed by maintenance imatinib.

DETAILED DESCRIPTION:
Induction therapy:

* Imatinib 200-400 mg p.o. daily x 10 days, Days 1-10 (see dose escalation scheme in Section 5.4 below).
* Mitoxantrone 10 mg/m2 daily x 5 days, Days 4-8.
* Etoposide 100 mg/m2 daily x 5 days, Days 4-8.
* Cytarabine 1.5 grams/m2 q12h x 4 doses, Days 9-10 (for patients aged 60 years and over, 1.0 gram/m2).

Only one induction course will be permitted. Only patients achieving CR will proceed to consolidation and maintenance.

Consolidation therapy, maximum 2 cycles (for patients achieving CR):

* Imatinib 200-400 mg p.o. daily x 8 days, Days 1-8 (see dose escalation scheme in Section 5.4 below).
* Mitoxantrone 12 mg/m2 daily x 2 days, Days 4-5.
* Cytarabine 3 grams/m2 q12h x 6 doses, Days 4,6,8. For patients aged 60 years and over, the dose will be reduced to 1.5 grams/m2.

Maintenance therapy (for patients still in CR at end of consolidation):

Imatinib 600 mg p.o. daily, until relapse or toxicity (see dose modification criteria in Section 5.6.6 below). Patients must receive at least one consolidation cycle before being permitted to proceed to maintenance therapy (see Section 5.6 for details). Maintenance therapy with imatinib will be provided for a maximum period of 1 year.

Dose escalation scheme:

Imatinib will be used during induction and consolidation at one of the following dose levels:

Level -1 100 mg daily Level 1 200 mg daily Level 2 300 mg daily Level 3 400 mg daily

ELIGIBILITY:
Inclusion Criteria:

* AML, all subtypes except APL.
* Prior induction therapy consisting of cytarabine 100-200 mg/m2 plus an anthracycline.
* One of the following:

  * persistent leukemia after induction therapy.
  * relapse within two years of achieving complete remission with induction therapy. Any consolidation therapy is acceptable, including stem cell transplantation.
* At least 10% bone marrow blasts, or biopsy confirmed extramedullary disease.
* Positivity for c-kit (CD117) in at least 30% of blasts as measured by flow cytometry.
* Aged 18-65.
* ECOG performance status < 3 (see Appendix I).
* No chemotherapy within the previous four weeks, other than hydroxyurea to control counts. If hydroxyurea is used, it must be stopped at least 24 hours prior to starting imatinib.
* Able to given informed consent.

Exclusion Criteria:

* Active uncontrolled infection.
* Active CNS leukemia.
* Serum creatinine > 200 umol/L.
* Serum bilirubin > 1.5 x ULN, AST or ALT > 2x ULN.
* Left ventricular ejection fraction < 50%.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2004-07; Primary Completion 2009-09 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Toxicity (hematologic and non-hematologic) of the combination of Imatinib and Chemotherapy consisting of Mitoxantrone, Etoposide and Ara-c | 2 years
  Hematologic toxicity
  * Number of days to ANC > 0.5 and 1.0.
  * Number of days until platelets > 20 and > 50, independent of platelet transfusions.
  * Number of days until RBC transfusion independent. Non-hematologic toxicity, as per NCI common toxicity criteria Hematologic dose-limiting toxicity (DLT) defined as > 40 days to ANC > 0.5 or platelets > 20 independent of transfusions.
Response rate - CR, MLFS and PR as per section 7.1 | 2 years
  * Complete response
  * Morphologic leukemia-free state
  * Partial remission (PR•No response (NR): Does not meet the criteria for CR, MLFS or PR.
Maximum tolerated dose of Imatinib when given in combination with chemotherapy | 2 years
  Maximum tolerated dose (MTD) of Imatinib (200, 300, 400 mg) when used in combination with NOVE-HiDAC induction and consolidation. MTD defined as highest dose resulting in up to 2/6 grade III-IV hematologic (as defined above) or non-hematologic DLTs per dose level. Non-hematologic DLTs as defined by NCIC CTC.

SECONDARY OUTCOMES:
Toxicity of imatinib maintenance therapy. | 2 years
  Hematologic
  * Number of days to ANC > 0.5 and 1.0.
  * Number of days until platelets > 20 and > 50, independent of platelet transfusions.
  * Number of days until RBC transfusion independent. Non-hematologic toxicity, as per NCI common toxicity criteria
Number of Participants with adverse events as a measure of safety and tolerability | 2 years
  Toxicity of imatinib maintenance therapy.
Remission-free survival and overall survival. | 2 years
  Median duration of remission free survival. Median overall survival and 2 year overall survival.
Total and phosphorylated c-kit activity at Days 1 and 4. | 2 years
  levels of total and phosphorylated c-kit - pre and post imatinib/Gleevec
Levels of downstream components of c-kit pathway at Days 1 & 4. | 2 years
  levels of phosphorylation ERK and AKT - pre and post imatinib/Gleevec

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada